CLINICAL TRIAL: NCT06855862
Title: An Exploration of the Relationship Between Serum Cytokine Levels and the Clinical Efficacy of Vedolizumab
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-207
Record Dates: First submitted 2025-02-24; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- clinical remission group: partial Mayo score ≤2 points and no subscore >1 point at week 16
- non-clinical remission group: partial Mayo score >2 points at week 16

SUMMARY:
It is uncertain the relationship between serum cytokine levels and the clinical efficacy of vedolizumab in the treatment of ulcerative colitis. The effects of cytokines on the efficacy of vidrecizumab in Chinese UC patients were retrospectively analyzed. Methods: Patients with UC were recorded. These patients were detected the levels of cytokines.

ELIGIBILITY:
Inclusion Criteria:

* UC patients Treated with Vedolizumab

Exclusion Criteria:

* pregnant
* had cognitive/developmental disorders that affected their ability to complete the study procedures
* had medical illness or therapies potentially affecting bone, nutrition or growth status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese ulcerative colitis treated with Vedolizumab
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
The partial Mayo score was applied to evaluate the clinical activity UC patients | 16 week and 34 week

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No